CLINICAL TRIAL: NCT01900093
Title: An Open-Label Prospective Proof-Of-Concept Trial to Evaluate the Response to Acthar Gel Therapy in Patients With Multiple Sclerosis (MS) Relapses Who Have Failed To Make an Adequate Recovery After Treatment With High-Dose Intravenous Methylprednisolone
Brief Title: Evaluation of the Response to Acthar Gel Therapy in Patients Who Failed Intravenous Methylprednisolone (IVMP) for MS Relapses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aaron Miller (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Aaron Miller, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-0600
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acthar Gel (Experimental): 80 units of subcutaneous Acthar Gel therapy daily
  Interventions: Drug: Acthar Gel

INTERVENTIONS:
Drug: Acthar Gel — 80 units of subcutaneous Acthar Gel therapy daily
  Other Names: Repository corticotrophin injection

SUMMARY:
Although ACTHAR gel is approved for the treatment of acute relapses, it is currently not widely used. Thus, we propose to conduct a small open-label proof-of-concept trial to evaluate the response to ACTHAR gel therapy in patients who have failed to make a satisfactory recovery after treatment with high dose IVMP. Documentation of the clinical course as well as any adverse events related to IVMP use will be made. The investigators propose to study the potential benefit of a 14-day course (the dose historically used since the landmark clinical trial of Rose et al1) of subcutaneous ACTHAR gel in 10 patients who have demonstrated inadequate improvement after a course of IVMP, 1000 mg daily, for 5 treatments (over a maximum of 8 days). These would be patients for whom PLEX would be considered as a treatment possibility. The primary outcome measure will be improvement in the targeted neurological deficit, as measured on the appropriate functional system score (FSS) of the EDSS.

DETAILED DESCRIPTION:
This is an open-label, small, proof-of-concept study examining the safety, tolerability, and extent of recovery of a two-week course of subcutaneous Acthar Gel therapy in patients with MS relapse who have failed to make a satisfactory recovery after treatment with high dose methylprednisolone. Eligible patients will be given 80 units of Acthar for 14 days. Patients will be evaluated at baseline, at 1 week of Acthar treatment, at completion of Acthar treatment, and 1 week after completion of treatment. For those who do not undergo plasmapheresis an additional evaluation will be conducted 2 weeks after completion of treatment. Monitoring will include blood pressure determination and blood sugar determination.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* EDSS of 2.0 - 7.5 (inclusive)
* Sustained a significant MS exacerbation affecting vision, brainstem, motor, or cerebellar function AND were initially treated with a 5 day course of IVMP within 10 days of the onset of symptoms.
* Failed to make adequate improvement and must initiate Acthar Gel therapy within two weeks (+/- 72 hours) after the first day of 5 treatments with 1000 mg IVMP, as judged by their treating neurologist.
* Must be able to comply with the requirements of the protocol as determined by the investigator.
* Ability to understand the purpose and risks of the study and provide signed and date informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.

Exclusion Criteria:

* Patients whose relapse consists of pure sensory or bowel/bladder symptoms
* History of ACTHAR gel use or other forms of ACTH with failure to improve or with occurrence of significant adverse experiences.
* Diagnosis of scleroderma, systemic fungal infections, ocular herpes simplex, congestive heart failure, and/or uncontrolled hypertension, and/or any clinically relevant medical disease that would put the patient at risk by participating in the study
* Persistent significant or severe infection
* Recent history of drug or alcohol abuse
* Concomitant use or prior use in the preceding 6 months of any investigational drug.
* Pregnant or nursing
* Recent surgery (up to the investigator's discretion what constitutes recent)
* History of, or the presence of, a peptic ulcer
* Known sensitivity to proteins of porcine origin
* Received a live or live attenuated vaccine in the last 30 days before baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in Functional System Score appropriate to the Targeted Neurological Deficit | at one week
  Primary outcome measure will be the percentage of patients improving by at least 1 step on the FSS appropriate to their neurological deficit (targeted neurological deficit [TND]} at 1 week following completion of treatment

SECONDARY OUTCOMES:
Improvement in Expanded Disability Status Scale | baseline and at 1 week
  Secondary outcome measures will be improvement in TND at completion of ACTHAR Gel therapy, improvement by at least 1 step on EDSS at completion of treatment and at 1 week following completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Miller, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Fred Lublin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Stephen Krieger, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Michelle Fabian, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Ilana Katz-Sand, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Sylvia Klineova, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Gretchen Mathewson, NP, Principal Investigator — Icahn School of Medicine at Mount Sinai; Aliza Ben-Zacharia, NP, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States